CLINICAL TRIAL: NCT04958018
Title: Influence of Almond Supplementation on Energy, Performance, and Inflammation Resolution From Exercise-Induced Muscle Damage
Brief Title: Almond Supplementation and Exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0102
Record Dates: First submitted 2021-06-17; First posted 2021-07-12 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Muscular Injury
Keywords: almonds; exercise; inflammation; oxylipins; cytokines
MeSH Terms: conditions — Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond (Experimental): 57 g almonds each day in split doses (half in the morning, half in the afternoon)
  Interventions: Dietary Supplement: Almonds
- Snack Bar (Active Comparator): snack bar group will ingest a matched calorie, common snack bar in split doses (324 calories/day, Nutri-Grain cereal bars, 120 kcal each)
  Interventions: Dietary Supplement: Snack bars

INTERVENTIONS:
Dietary Supplement: Almonds — almond (Prunus dulcis) consumption
  Arms: Almond
Dietary Supplement: Snack bars — 324 calories/day, Nutri-Grain cereal bars, 120 kcal each
  Arms: Snack Bar

SUMMARY:
The PURPOSE of this study is to see if eating almonds for four weeks will reduce muscle damage, soreness, and inflammation during several days of recovery from eccentric exercise.

DETAILED DESCRIPTION:
This will be the first study to determine if 4-weeks ingestion of nutrient-dense almonds improves feelings of energy and vitality, and mitigates post-exercise inflammation (plasma cytokine and oxylipin levels), muscle soreness, and muscle damage. An acute 90-minute bout of eccentric exercise will be used to induce muscle damage and inflammation in a group of 60 relatively untrained male and female adults (ages 30-65 years). Using a randomized, parallel group design, almond supplementation (57 g/d) for a 4-week period prior to the eccentric exercise challenge will be investigated as a countermeasure strategy to exercise-induced muscle damage and inflammation. The control group will ingest a calorie-matched common snack (cereal bars). To improve the potential for capturing an intervention effect, advanced mass spectrometry procedures will be utilized to measure changes in 70 different oxylipins and lipid mediators that are involved in regulating inflammation. C-reactive protein (CRP), six inflammatory cytokines, and muscle damage biomarkers will also be measured. Blood samples (7 total) will be collected before and after the 4-week supplementation period, and then daily during 5 days of recovery from the eccentric exercise bout. The Profile of Mood States (POMS) will be used to measure mood state and specific domains including vigor or activity, and fatigue or inertia. Exercise performance will be measured each time a blood sample is collected using a comprehensive battery that includes vertical jump, leg/back muscle strength, bench press muscle endurance, and anaerobic power (30-second Wingate test).

Participants will be randomized to the almond or typical snack (cereal bars) supplement groups. The parallel group design is being utilized in this study because of the "repeat exercise bout" effect (i.e., post-exercise muscle damage and inflammation are reduced when the same bout is repeated within days and weeks of the first bout). Participants will come to the lab at 7:00 am at the beginning of the 4-week supplementation period, and then Monday (eccentric exercise bout) and Tuesday through Friday (recovery) in an overnight fasted state. The 4-week supplementation period was based on practical issues related to the research design. A 4-week almond supplementation period was commonly used in prior studies and was sufficient to demonstrate favorable blood lipid changes relative to control conditions.

Seven blood samples will be collected and analyzed for various measures of muscle damage, oxylipins, and inflammation. After each of the blood draws, participants will complete the POMS (energy, vitality) and provide a muscle soreness rating (DOMS). Physical activity will be monitored during the entire study using the International Physical Activity Questionnaire (IPAQ). The IPAQ was developed to measure health-related physical activity (PA) in populations. The short version of the IPAQ has been tested extensively and is now used in many international studies.

Study participants will come to the performance lab for orientation to the testing procedures. This will include a review of the consent form, completion of basic questionnaires, and an introduction to the eccentric muscle exercise bout and the strength/power performance testing protocol (about 1.5 hours) (visit #1). This will be followed by another lab session for pre-study measurements and sample collection with subjects in an overnight fasted state (visit #2) (see description below). A 3-day food record will be collected during the end of the 4-week supplementation period to assess the background diet.

Study participants will have to agree to 5 other lab visits during a one-week period (all overnight fasted condition). These lab visits will start at 7:00 am on Monday, with morning visits at 7:00 am on Tuesday through Friday. At each of the 5 lab visits, study participants will come to the lab at 7:00 am not having consumed food or beverages (other than water) for at least the previous 9 hours, and having abstained from vigorous exercise for at least the previous 24-48 hours. The Monday session will take about 2.5 hours (7:00 to 9:30 am), and the Tuesday through Friday sessions will take about 30-45 minutes each. The total amount of time participants will be asked to volunteer for this study is about 8-9 hours at the performance lab.

Participants will be randomized to almond or snack groups, and provided a 4-weeks supply of supplements. Participants in the almond group will consume 57 g almonds each day in split doses (half in the morning, half in the afternoon). Participants in the snack group will ingest a matched calorie, common snack bar in split doses (324 calories/day, Nutri-Grain cereal bars, 120 kcal each).

The daily dose of almonds (57 g) and just under 3 Nutri-Grain cereal bars will provide a distinct difference in nutrient intake. A serving of 57 g of almonds has 324 calories with 12 g of protein, 28 g of fat (17 g from monounsaturated, 6.6 g from polyunsaturated, 2.6 g from saturated), 12 g of carbohydrates and 6.6 g of fiber, 160 mg total polyphenols, and significant amounts of vitamin E (96% RDA), magnesium, manganese, copper, and other minerals.

Baseline Testing (Visit #2) Participants will provide a blood sample using standard phlebotomy procedures. Participants will also provide a spot urine sample, with instructions to capture a mid-stream urine sample in a disposable urine cup. Spot urine samples provide valid metabolite data as indicators of dietary intake. Height, body weight, and body composition will be measured in a private section of the lab. Bioelectrical impedance (BIA) using the seca BIA scale will be used to assess body composition (i.e., the percent of body weight that is fat tissue) and body weight. Participants will remove shoes and socks and stand with bare feet on the seca scale for about 7-10 seconds while grasping side rails with your hands. Percent body fat will also be measured using the BodPod. Participants will sit inside the BodPod with a tight-fitting swim suit for about 10 minutes while body fat is calculated. The Profile of Mood States (POMS) will be administered. Delayed onset of muscle soreness (DOMS) will be assessed using a 1-10 scale.

Participants will perform some light exercises to warm up, followed by five muscle function tests: vertical jump, bench press, leg-back strength, 60-yard shuttle run test, and anaerobic power through the 30-second Wingate test.

1. Vertical jump: Participants will first stand erect with the feet flat on the floor and reach as high as possible with both arms and hands (standing reach height). Participants will then squat down and jump as high as possible with one arm and hand, and tap the measuring device on the Vertec vertical jump apparatus (jump height). This will be repeated three times, with the best score recorded as the difference between the jump and standing reach heights.
2. Bench press to exhaustion at 50%/75%: Participants will lie down supine on a bench, and with spotters standing on either side attempt to bench press a weighted bar equal to 75% (males) or 50% (females) body weight as many times as possible (to a metronome set at 60 beats/min or 30 lifts/min). The bar must touch a foam block on the chest lightly in the down position, and the arms must be straight in the up position.
3. Leg-Back Strength: Leg/lower back strength will be assessed with a dynamometer. With the legs slightly bent at the knee, participants will grasp a bar attached via a chain and a force measuring device with straight arms, and then lift up with maximal effort for several seconds. This will measure the isometric strength of both legs and back, and will be repeated three times.
4. 30-Second Wingate Cycling Test, Anaerobic Power: The Lode cycle ergometer will be adjusted to the participant's body weight (7 watts per kilogram). After a warm up, participants will sprint cycle at maximal speed for 30 seconds. The peak power and average power will be recorded and adjusted to body weight.
5. 60-Yard Shuttle Run Test: The shuttle run is a test of anaerobic speed endurance and agility, in which participants run to 5 yards, 10 yards, 15 yards, there and back, for a total of 60 yards. This is a ladder shuttle of progressing distances. Four marker cones are placed 5 yards apart. The participant starts from one end, runs 5 yards and back to the start, 10 yards and back, then 15 yards and finishes at the start line. A total of 60 yards is completed. The participant is required to touch the line with their hand at each turn, and runs through the finish line, for a total of five touches. The time to complete the test in seconds is recorded. The score is the best time of three trials.

Testing Sequence, Day of Eccentric Muscle Exercise (Monday) and 4-Days Recovery (Tuesday through Friday):

Participants will come to the lab at 7:00 am in an overnight fasted state (i.e., no food or beverages other than water for at least the previous 9 hours). Participants (on Monday only) will provide a spot urine sample that will be aliquoted, stored in a -80°C freezer, and then sent to Metabolon (Durham, NC) for global metabolomics analysis (to capture metabolite shifts related to almond ingestion). Participants will provide a blood sample, fill in the POMS, and give a DOMS rating. The almond or snack supplements (half dose) will be consumed. Participants will perform some light exercises to warm up, followed by five muscle function tests (same as baseline): vertical jump, bench press, leg-back strength, 60-yard shuttle run test, and anaerobic power through the 30-second Wingate test. Participants will take these performance tests before and after the 90-minute eccentric muscle exercise bout, and each of the following four mornings at the performance lab.

After taking the five performance tests, participants will engage in 90-minutes of eccentric exercise. This protocol induces significant muscle damage and soreness.

Immediately following exercise, participants will provide a muscle soreness rating and a blood sample. Participants will then take the five muscle function tests. Participants will ingest the supplements (half-dose) during the afternoon. Participants will return at 7:00 am in an overnight fasted state four days in a row (Tuesday through Friday) after Monday's eccentric exercise bout, and provide muscle soreness ratings and blood samples followed by ingestion of the supplements (half dose). Following ingestion of the supplements, participants will take the five muscle function tests. Participants will the second half dose of the supplements in the afternoon (Tuesday, Wednesday, Thursday). On Friday morning, participants will take the supplement (half dose) prior to the muscle function tests. During this week of testing, participants will engage in normal training.

The blood and urine samples will be analyzed for a panel of oxylipins, CRP and six cytokines, three muscle damage markers (creatine kinase, myoglobin, LDH), and urine metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 30-65 years.
* Non-smoker.
* Body mass index of 23 to 30 kg/m2.
* Not engaged in regular weight lifting (less than 3 sessions per week).
* Agree to train normally, maintain weight, and avoid the regular use of protein supplements, large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation (especially Advil, Motrin, aspirin, and similar drugs) during the study.
* Categorized as "low risk" using a screening questionnaire.
* Generally healthy and without disease including heart disease, stroke, cancer, diabetes, arthritis.
* Willing to collect two 24-hour urine samples.

Exclusion Criteria:

* Inability to comply with study requirements.
* Engaged in regular weight training (3 or more times a week).
* Pregnant or breastfeeding.
* Any other condition that would interfere with successful completion of the study.
* Current diagnosis of heart disease, diabetes, or cancer (except for skin cancer).
* History of allergic reactions to almonds or cereal bars.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Serum concentration of creatine kinase | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle damage biomarker

SECONDARY OUTCOMES:
Plasma concentrations of pro-inflammatory oxylipins: 19-hydroxy-eicosatetraenoic acid (HETE), 20-HETE, 20-cooh-AA, 8,9-dihydroxy-eicosatrienoic (all ng/ml) acid; (diHETrE), 14,15-diHETrE | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Inflammation biomarkers
Plasma concentration of IL-6 | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Inflammation biomarkers
Urine almond metabolites: epicatechin, catechin, epiafzelechin, gallic acid, ellagic acid (all uM) | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Almond polyphenol gut-derived metabolites
30-second Wingate cycle test watts | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Anaerobic sprint power cycling test, peak and average watts
Leg-back strength kilograms | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle performance, leg-back strength with a dynamometer
Bench press repetitions | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle performance, bench press to exhaustion with weighted bar
Vertical jump height | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Vertical jump height as a muscle function test
Rating of Profile of Mood States (POMS) | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Rating scale to assess mood states, energy, vitality; 0 to 4 scale, with 0=not at all and 4 = extremely
Serum concentration of myoglobin | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle damage biomarker

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will provide data upon request.